CLINICAL TRIAL: NCT05031767
Title: Remote Monitoring of Axial Spondyloarthritis in Specialist Healthcare Services
Brief Title: Remote Monitoring of Axial Spondyloarthritis
Acronym: ReMonit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diakonhjemmet Hospital (Other)
Responsible Party: Principal Investigator, Nina Osteras, Principal investigator, Diakonhjemmet Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: REK no.:229187
Record Dates: First submitted 2021-08-23; First posted 2021-09-02 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Axial Spondyloarthritis
Keywords: rheumatic diseases; musculoskeletal diseases; joint diseases; arthritis
MeSH Terms: conditions — Axial Spondyloarthritis; Rheumatic Diseases; Musculoskeletal Diseases; Joint Diseases; Arthritis | interventions — Remote Patient Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual care (Active Comparator): Conventional current follow-up strategy
  Interventions: Other: Usual care
- Remote monitoring (Experimental): Remote monitoring by health professionals at the hospital
  Interventions: Other: Remote monitoring
- Patient-initiated care (Experimental): No pre-scheduled visits or remote monitoring.
  Interventions: Other: Patient-initiated care

INTERVENTIONS:
Other: Usual care — Conventional follow-up strategy with blood tests, patient-reported outcomes, and pre-scheduled visits at the hospital every 6th month.
  Continue using medical treatment with tumour necrosis factor inhibitors (TNFi). Patients will be instructed to use NSAIDs should they experience minor worsening of symptoms, but if the patients experience significant symptom worsening and suspect a severe disease worsening (flare) or adverse events, they will be instructed contact the hospital.
  Arms: Usual care
Other: Remote monitoring — Hospital health professionals perform remote monitoring of frequent patient-reported outcomes, blood test results, and physical activity data available on a digital platform.
  Continue using medical treatment with tumour necrosis factor inhibitors (TNFi). Patients will be instructed to use NSAIDs should they experience minor worsening of symptoms, but if the patients experience significant symptom worsening and suspect a severe disease worsening (flare) or adverse events, they will be instructed contact the hospital .
  Arms: Remote monitoring
Other: Patient-initiated care — No pre-scheduled visits or remote monitoring.
  Continue using medical treatment with tumour necrosis factor inhibitors (TNFi). Patients will be instructed to use NSAIDs should they experience minor worsening of symptoms, but if the patients experience significant symptom worsening and suspect a severe disease worsening (flare) or adverse events, they will be instructed contact the hospital.
  Arms: Patient-initiated care

SUMMARY:
The ReMonit study is a 18-months, non-inferiority randomized, controlled trial with three parallel arms to determine if two, new follow-up strategies for patients with axial spondyloarthritis (axSpA) are non-inferior in maintaining stable, low disease activity over time compared to the conventional follow-up regimen with regular hospital visits.

DETAILED DESCRIPTION:
The trial will include Norwegian adult males and females with axial spondyloarthritis.

240 participants will be randomized 1:1:1 to either:

1. Control group: a. Usual care, i.e. conventional follow-up strategy with blood tests, patient-reported outcomes (PROs), and pre-scheduled visits at the hospital every 6th month
2. Remote monitoring: hospital health professionals (HPs) perform remote monitoring of frequent PROs, blood test results, and physical activity data available on a digital platform
3. Patient-initiated care: no pre-scheduled visits or remote monitoring

The study has 18 months follow-up. We will use a 15% non-inferiority margin.

The study will also include qualitative research including semi-structured interviews and observations of patients in the two intervention groups and health professionals involved in the study. The interviews will explore experiences with remote monitoring and video consultations.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-nursing female >18 years of age at screening
* Patients with a diagnosis of axSpA who fulfil the diagnostic Assessment of SpondyloArthritis International Society (ASAS) criteria for axSpA
* Stable medical treatment with TNFi the last 6 months
* Low disease activity (ASDAS<2.1) at inclusion
* Capable of understanding the Norwegian language and of signing an informed consent form

Exclusion Criteria:

Medical conditions:

* Major co-morbidities, such as severe malignancies, severe diabetes mellitus, severe infections, uncontrollable hypertension, severe cardiovascular disease (NYHA class III or IV), severe respiratory diseases, and/or cirrhosis.
* Indications of active tuberculosis (TB)

Diagnostic assessments:

* Abnormal renal function, defined as serum creatinine >142 µmol/L in female and >168 µmol/L in male, or glomerular filtration rate (GFR) <40 mL/min/1.73 m2
* Abnormal liver function (defined as Alanine Transaminase (ALT) >3x upper normal limit), active or recent hepatitis
* Leukopenia and/or thrombocytopenia

Other:

* Pregnancy and/or breastfeeding (current at screening or planned within the duration of the study)
* Severe psychiatric or mental disorders, alcohol abuse or other substance abuse, language barriers or other factors which makes adherence to the study protocol impossible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2021-09-07 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Low disease activity at follow-up | 6 months
  The proportion of patients with low disease activity (defined as ASDAS <2.1) at the 6-months follow-up
Low disease activity at follow-up | 12 months
  The proportion of patients with low disease activity (defined as ASDAS <2.1) at the 12- months follow-up
Low disease activity at follow-up | 18 months
  The proportion of patients with low disease activity (defined as ASDAS <2.1) at the 18-months follow-up

SECONDARY OUTCOMES:
Ankylosing Spondylitis Disease Activity Score (ASDAS) | Baseline, 6, 12 and 18 months
  Ankylosing Spondylitis Disease Activity Score (ASDAS) is a clinical measure of disease activity calculated from four patient-reported outcomes (PROs) and C-reactive Protein (CRP) (or erythrocyte sedimentation rate (ESR) if CRP is not available). The formula for calculating ASDAS CRP = 0.12 × back pain + 0.06 × duration of morning stiffness + 0.11 × patient global + 0.07 × peripheral pain/swelling + 0.58×Ln(CRP + 1)). Higher values indicate worse outcome.
Ankylosing Spondylitis Disease Activity Score (ASDAS) | Every month, maximum 18 months
  Monthly for a subgroup among the Remote monitoring group. ASDAS is a clinical measure of disease activity calculated from four PROs and CRP (or ESR if CRP is not available). The formula for calculating ASDAS CRP = 0.12 × back pain + 0.06 × duration of morning stiffness + 0.11 × patient global + 0.07 × peripheral pain/swelling + 0.58×Ln(CRP + 1)). Higher values indicate worse outcome.
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | Baseline, 6, 12 and 18 months
  Patient-reported disease activity last 7 days on 6 items using a numeric rating scale (NRS) 0-10. The score is the sum (of the first four individual questions and the mean of questions five and six) divided by five. The sum score range 0-10; higher value indicate worse outcome.
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | Every month, maximum 18 months
  Monthly reported by the Remote monitoring group if disease worsening. Patient-reported disease activity last 7 days on 6 items using a NRS 0-10. The score is the sum (of the first four individual questions and the mean of questions five and six) divided by five. The sum score range 0-10; higher value indicate worse outcome.
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | Baseline, 3, 6, 9, 12, 15 and 18 months
  Reported every third month by the Patient-initiated care group if disease worsening. Patient-reported disease activity last 7 days on 6 items using a NRS 0-10. The score is the sum (of the first four individual questions and the mean of questions five and six) divided by five. The sum score range 0-10; higher value indicate worse outcome.
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | Every month, maximum 18 months
  Reported monthly by the a subgroup among the Remote monitoring group. Patient-reported disease activity last 7 days on 6 items using a NRS 0-10. The score is the sum (of the first four individual questions and the mean of questions five and six) divided by five. The sum score range 0-10; higher value indicate worse outcome.
C-Reactive Protein (CRP) | Every month, maximum 18 months
  CRP measured at home in a subgroup among the Remote monitoring group
Patient global assessment of disease activity | Baseline, 6, 12 and 18 months
  Patient-reported disease activity last 7 days on a NRS 0-10 ; higher value indicate worse outcome
Patient global assessment of disease activity | Every month, maximum 18 months
  Monthly reported by the Remote monitoring group. Patient-reported disease activity last 7 days on a NRS 0-10 ; higher value indicate worse outcome
Patient global assessment of disease activity | 3, 6, 9, 12, 15 and 18 months
  Reported every third month by the Patient-initiated care group: Patient-reported disease activity last 7 days on a NRS 0-10 ; higher value indicate worse outcome
Patient-reported flare | 6, 12 and 18 months
  Patient-reported experience of a significant worsening of symptoms (reflecting a flare in disease activity), response options: no, yes, uncertain. If yes or uncertain, they will be asked which date the flare occurred and the number of days it lasted.
Patient-reported flare | Every month, maximum 18 months
  Monthly reported by the Remote monitoring group. Patient-reported experience of a significant worsening of symptoms (reflecting a flare in disease activity), response options: no, yes, uncertain. If yes or uncertain, they will be asked which date the flare occurred and the number of days it lasted.
Patient-reported flare | 3, 6, 9, 12, 15 and 18 months
  Reported every third month by the Patient-initiated care group. Patient-reported experience of a significant worsening of symptoms (reflecting a flare in disease activity), response options: no, yes, uncertain. If yes or uncertain, they will be asked which date the flare occurred and the number of days it lasted.
Bath Ankylosing Spondylitis Functional Index (BASFI) | Baseline, 6, 12 and 18 months
  10 item questionnaire (NRS 0-10) used to assess disease activity last 7 days. The score is the sum of each individual question divided by 10, higher value indicate worse outcome.
Activity Impairment | Baseline, 6, 12 and 18 months
  Item no.6 from Work Productivity and Activity Impairment (WPAI): self-reported activity impairment on a NRS 0-10; higher value indicate worse outcome.
Patient-reported global change in disease activity | 6, 12 and 18 months
  Single item with seven-point response scale ranging from "Much worse" to "Much better".
Patient-reported global change in activity impairment | 6, 12 and 18 months
  Single item with seven-point response scale ranging from "Much worse" to "Much better".
Pain (general) | Baseline, 6, 12 and 18 months
  Self-reported pain level last 7 days hours on a NRS 0-10; higher value indicate worse outcome.
Joint pain | Baseline, 6, 12 and 18 months
  Self-reported joint pain level last 7 days hours on a NRS 0-10; higher value indicate worse outcome.
Sleep impairment | Baseline, 6, 12 and 18 months
  1 item from Pittsburgh Sleep Quality Index, self-reported sleep impairment in last month due to pain with 4 response categories ranging "Not during the past month" to "Three or more times a week" ; higher value indicate worse outcome.
Patient satisfaction with care | Baseline, 6, 12 and 18 months
  1 item with five point response options ranging from "Very satisfied" to "Very dissatisfied", higher value indicate better outcome
Daily steps | Through study completion, maximum 18 months
  Remote monitoring and Patient-initiated care groups, number of steps during daytime captured by wearing a smartwatch
Mean pulse level | Through study completion, maximum 18 months
  Remote monitoring and Patient-initiated care groups, mean pulse level during daytime captured by wearing a smartwatch
Euro Quality of Life 5 Dimensions 5 Levels (EQ5D-5L) | Baseline, 6, 12 and 18 months
  6 item utility instrument for measurement of health related quality of life, 5 first items with 5 response categories, item no.6: self-reported health status on a 0-100 mm scale
Concomitant medication | Baseline, 6, 12 and 18 months
  Self-reported use of NSAIDs and analgesics and national register data from The Norwegian Prescription Register
Swollen joint count | Baseline, 6, 12 and 18 months
  For the Control group, examiner assessed metacarpophalangeal (MCP) 1-5, proximal interphalangeal (PIP) 1-5, wrists, elbows, shoulders, ankles, forefeet
Swollen joint count | Baseline, through study completion, and 18 months
  At extra visits/withdrawals/early discontinuation in the Remote monitoring and Patient-initiated care groups, For the Control group, examiner assessed MCP 1-5, PIP 1-5, wrists, elbows, shoulders, ankles, forefeet
Tender joint count | Baseline, 6, 12 and 18 months
  For the Control group, examiner assessed MCP 1-5, PIP 1-5, wrists, elbows, shoulders, ankles, forefeet
Tender joint count | Baseline, through study completion, and 18 months
  At extra visits/withdrawals/early discontinuation in the Remote monitoring and Patient-initiated care groups, For the Control group, examiner assessed MCP1-5, PIP 1-5, wrists, elbows, shoulders, ankles, forefeet
Heel enthesitis | Baseline, 6, 12 and 18 months
  For the Control group, the presence of heel enthesitis is examined clinically by a health professional. Scored as not present/present right heel/present left heel/present both heels.
Heel enthesitis | Baseline, through study completion, and 18 months
  At extra visits/withdrawals/early discontinuation in the Remote monitoring and Patient-initiated care groups, , the presence of heel enthesitis is examined clinically by a health professional. Scored as not present/present right heel/present left heel/present both heels.
Costs related to hospital visits | Baseline
  Self-reported way of transport to the hospital; walking or bicycling/private car/public transportation/taxi/airplane/other.
Costs related to hospital visits | Baseline
  Self-reported travel distance in kilometres to the hospital.
The need to take time off work for hospital visits or video consultations | Baseline
  If in paid work, the need to take time off from work is indicated as yes or no.
Health care utilization | Baseline, 6, 12 and 18 months
  Self-reported health care use and national register data on consultations and treatment in secondary and primary health care
Extra visits, telephone and video consultations | Through study completion, maximum 18 months
  Number of extra visits to the hospital or video consultations with a health care provider
Withdrawals/Early discontinuation | Through study completion, maximum 18 months
  Number of withdrawals/early discontinuation
Adverse events | Through study completion, maximum 18 months
  Number of adverse events, serious adverse events, and withdrawals because of adverse events.
Patient-reported self-efficacy for using different digital devices, secure login and digital health services measured on a Likert scale | Baseline
  Self-efficacy/confidence in using smartphone, tablet, computer, app's, secure login and digital health services. 6 items with Likert scale response categories: Never used, Very bad, Bad, Neither good nor bad, Good, Very good. Score range 1-5; higher scores indicate higher self-efficacy.
eHealth literacy | Baseline
  20 items from 4 domains of the eHealth Literacy Questionnaire (eHLQ). Four point response scale, sum domain score range 1-4. Lower scores indicate lower eHealth literacy.
Body signs and symptoms | 18 months
  To what degree do you understand your body's signs and symptoms. Single item, 4-point Likert scale (not at all - to a large degree + do not know-option)
Patient satisfaction with remote monitoring or patient-initiated care | 18 months
  Service User Technology Acceptability Questionnaire (SUTAQ) reported by the Remote monitoring group. 22 items in 5 subscales. Score range 1-6. Higher scores in subscales 1,2 and 5/lower scores in subscales 3 and 4 indicate higher acceptability with telehealth.
Patient satisfaction with remote monitoring or patient-initiated care | 18 months
  Service User Technology Acceptability Questionnaire (SUTAQ) reported by the Patient-initiated care group. 3 of 22 items: #1, #10 and #11. Score range 1-6. Higher scores in indicate higher acceptability with telehealth.
Preferred follow-up strategy | 18 months
  One item on whether the preferred follow-up strategy would be Remote monitoring or Patient-initated care reported by the two intervention groups only.

CONTACTS AND LOCATIONS:
Overall Officials: Tore Kvien, MD, Professor em, Study Chair — Diakonhjemmet Hospital
Locations (1):
- Diakonhjemmet Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Berg IJ, Tveter AT, Bakland G, Hakim S, Kristianslund EK, Lillegraven S, Macfarlane GJ, Moholt E, Provan SA, Sexton J, Thomassen EE, De Thurah A, Gossec L, Haavardsholm EA, Osteras N. Follow-Up of Patients With Axial Spondyloarthritis in Specialist Health Care With Remote Monitoring and Self-Monitoring Compared With Regular Face-to-Face Follow-Up Visits (the ReMonit Study): Protocol for a Randomized, Controlled Open-Label Noninferiority Trial. JMIR Res Protoc. 2023 Dec 27;12:e52872. doi: 10.2196/52872. PMID 38150310

DOCUMENTS (1):
  • Study Protocol (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/67/NCT05031767/Prot_000.pdf